CLINICAL TRIAL: NCT02873312
Title: Prospective, Multi-Center, Randomized, Double-Blinded Trial of Percutaneous Tibial Nerve Stimulation With the Bioness StimRouter Neuromodulation System Versus Sham in the Treatment of Overactive Bladder (OAB)
Brief Title: Overactive Bladder Treatment Using StimRouter Neuromodulation System: A Prospective Randomized Trial
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Bioness Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CP-STMR-OAB-002
Record Dates: First submitted 2016-08-10; First posted 2016-08-19 (Estimated); Last update posted 2021-01-29 (Actual); Status verified 2020-07

CONDITIONS: Overactive Bladder
MeSH Terms: conditions — Urinary Bladder, Overactive

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: The implanting investigator, the study subjects, and the individuals who assess the outcome measures for each subject will be blinded to the subjects' randomization groups. Each study site's programmers will be unblinded to the randomization assignment and will receive each subject's randomization assignment. The programmers will then set the stimulation parameters and train the subjects on device use.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- StimRouter Treatment (Experimental): The Treatment group will receive therapeutic level StimRouter electrical stimulation. At the end of the Month 3 visit the Treatment group will continue to receive therapeutic level StimRouter electrical stimulation for an additional 3 months.
  Interventions: Device: StimRouter
- StimRouter Control (Sham Comparator): The Control group will receive sham (sub-therapeutic level only) StimRouter stimulation. At the end of the Month 3 visit the Control group will be allowed to receive therapeutic level StimRouter electrical stimulation for 3 months.
  Interventions: Device: StimRouter

INTERVENTIONS:
Device: StimRouter — The StimRouter System is a neuromodulation system consisting of the following components and accessories:
  * An implantable multi-electrode lead with integrated receiver in loader and surgical tools for implantation of the implantable lead.
  * An external programming system with a clinician programmer, a clinician programmer cradle and charger, an external pulse transmitter tester and accessories.
  * A patient-operated system with an external pulse transmitter (StimRouter EPT), a disposable StimRouter Electrode, an external patient programmer and charger, and accessories.
  Other Names: StimRouter Neuromodulation System

SUMMARY:
Approximately 20 Study Sites will participate over total 24 months. Study population will consist of adults age 22 or over, reporting overactive bladder (OAB) symptoms for at least 3 months.

Primary Study Objectives:

1. To assess efficacy of the StimRouter stimulation in improving OAB symptoms of urgency and frequency as measured by Patient Voiding Diary when targeting the posterior tibial nerve
2. To assess safety of the StimRouter therapy for the indication of OAB

Secondary Study Objective:

To evaluate efficacy of the StimRouter therapy in addressing urinary urge incontinence as measured by the Patient Voiding Diary

Study Design is prospective, multi-center, randomized, double-blinded

Primary Endpoint:

The primary efficacy endpoint will be the difference between the investigational and control groups in proportion of responders, where Responder is defined as having ≥50% improvement in average voiding frequency above the normal value of 8 (those returning to normal voiding based on 7-day average voids/leak episodes < 9, will be categorized as achieving half or more reduction) AND having ≥50% improvement in average number of moderate to severe urgency episodes, at approximately three months after programming.

Secondary Endpoint:

Secondary endpoint will be the difference between the investigational and control groups in proportion of patients with reduction by half or more in urinary urge incontinence as measured by the average number of urge incontinence episodes per day.

DETAILED DESCRIPTION:
Approximately 180 subjects will be enrolled in the Percutaneous Tibial Nerve Stimulation (PTNS) for Overactive Bladder study. After signing the informed consent and completing the screening visit, eligible candidates will be asked to (1) stop any OAB medications (including but not limited to anti-muscarinic medication or tricyclic antidepressants (TCA) as well as stabilize dosage and frequency of any concomitant medications for 3 weeks, if applicable, and then (2) complete a daily Patient Voiding Diary for 7 days .

Subjects will then return to the office for baseline review. If all screening and baseline criteria are met, the subject will be enrolled, randomized in a 1:1 ratio into either the "control group" or the "investigational group" and scheduled for implant with the StimRouter device.

After approximately 3 weeks for healing post-implant, study participants will be programmed according to their randomization assignment. All subjects will be instructed to apply stimulation at least 3 days/week for at least 30 minutes/day (i.e., the minimum protocol requirements for device use) for 6 months and to apply stimulation when they anticipate OAB events. Patient Voiding Diaries will be completed by the participants for 7 days prior to each follow-up visit and provided to the office at each follow-up visit. Follow-up visits will occur at Month 1, Month 2, Month 3, Month 5 and Month 6. Each follow-up visit will include the review of subject voiding diaries and the completion of other subject questionnaires for measuring OAB and quality of life assessments. Final follow-up evaluations for all subjects will occur at Month 6.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female age ≥22 years and competent to provide consent
2. Minimum 3 months of self-reported OAB symptoms
3. A mean score of ≥4.0 on the OAB-q symptom questions 1-8
4. Diagnosis of OAB with Overactive Bladder Symptom Score (OABSS) ≥ 8.0
5. Average urinary frequency of ≥ 10 daily voids associated with urgency
6. Able to tolerate and sense tibial nerve stimulation
7. Willing to discontinue OAB and/or tricyclic antidepressant (TCA) medications for 3 weeks prior to the implant and for the entire study period and not to change dosages/frequency of all others for 3 weeks prior to the implant
8. Failed/inadequate response to first- and second-line therapy for OAB
9. Body mass index (BMI) < 31 or investigator does not expect BMI to interfere with ability to place the implant or negatively impact healing at implant site
10. Able to toilet self and have and maintain good personal hygiene
11. Able to utilize the StimRouter system independently
12. Negative urine dipstick result (no UTI detected)
13. If female of child-bearing age, willing to use a medically-acceptable method of contraception for the duration of the study (e.g. oral contraceptives, condoms, shot, patch, etc.)
14. Able to provide clear, thoughtful responses to questions and questionnaires
15. Willing to visit office for device programming and clinical evaluations at 1, 2, 3, 5 and 6 months after starting external device usage
16. Willing to complete a Patient Voiding Diary for 7 consecutive days prior to implant and 7 consecutive days before each follow-up visit, with moderate to severe urge component at Baseline

Exclusion Criteria:

1. Neurogenic bladder
2. Urinary tract mechanical obstruction including but not limited to Benign Prostatic Hyperplasia (BPH), treated or untreated, with ongoing significant obstruction
3. Treatment of bladder or pelvic floor dysfunction with botulinum toxin (Botox ®) or surgery in past 12 months
4. Urinary tract, bladder or vaginal infection or inflammation
5. More than minimal level of stress incontinence or mixed incontinence with stress component likely to confound study outcome
6. Type I diabetes or uncontrolled Type II diabetes
7. Allergy to local anesthetic or adhesives
8. Bleeding disorder or on an anticoagulant that cannot be stopped for 3 days before the implant
9. Pregnant, lactating, planning to become pregnant, given birth in the past 12 months, or female of child-bearing potential and not practicing a medically-approved method of birth control
10. Skin lesions or compromised skin at the implant or stimulation site
11. Use of investigational drug or device therapy or participation in any study involving or impacting gynecologic, urinary or renal function within past 4 weeks
12. Implanted neurostimulator, pacemaker, or defibrillator
13. Current use of TENS in pelvic region, back or leg
14. Current or prior use of electrical stimulation therapy for OAB (e.g. PTNS, sacral nerve stimulation, pelvic floor muscle stimulation or biofeedback)
15. Metallic implant below knee, within 6 inches of proposed site for implanted lead
16. Prior vaginal mesh or similar surgery that has not abolished stress incontinence, intravaginal pessaries, or other evidence of stress incontinence significant enough to confound study
17. Requirement for serial MRIs
18. Presence of a documented condition or abnormality that could compromise the safety of the patient
19. Life expectancy of less than 1 year

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2017-02-10 (Actual); Primary Completion 2021-07-30 (Estimated); Study Completion 2021-07-30 (Estimated)

PRIMARY OUTCOMES:
1) Patient Voiding Diary | Baseline, Month 3
  The daily Patient Voiding Diary is a self-reported record and it includes how frequently the patient intentionally urinates during the day (frequency) and is awakened to urinate at night (nighttime void frequency), amount voided, number of urgency episodes, voids with moderate to severe urgency, urinary urge incontinence episodes and the degree of urgency to urinate. The 7-day daily Patient Voiding Diary will be assessed at baseline and at approximately 3 months after programming to measure total number of voids (frequency) and voids with moderate-to-severe urgency.The average for each of the seven-day periods will be calculated and compared.
Adverse Events reported cumulatively throughout study | Baseline through Month 6
  Occurrence of anticipated and unanticipated adverse events will be documented, accumulated and reported for the duration of the study

SECONDARY OUTCOMES:
Seven-Day Patient Voiding Diary | Baseline, Month 3
  The 7-day daily Patient Voiding Diary will be assessed at baseline and at approximately 3 months after programming to measure urinary urge incontinence episodes.

CONTACTS AND LOCATIONS:
Overall Officials: Keith McBride, Study Chair — Bioness Inc; Howard Goldman, MD, Principal Investigator — The Cleveland Clinic
Locations (19):
- United States (15):
  - Del Sol Research, Tucson, Arizona
  - Kaiser Permanente Reserach, Irvine, California
  - University of Southern California, Los Angeles, California
  - Providence St. John's Health Center, Santa Monica, California
  - Skyline Urology, Sherman Oaks, California
  - Barrett Cowan, MD, Urology Associates, Englewood, Colorado
  - Clinical Research Center of Florida, Pompano Beach, Florida
  - Meridian Clinical Research, LLC/Urology Associates Savannah, Savannah, Georgia
  - Comprehensive Urologic Care, Barrington, Illinois
  - Sheldon Freedman, MD LTD, Las Vegas, Nevada
  - University of North Carolina Urogynecology, Chapel Hill, North Carolina
  - Cleveland Clinic Glickman Urologic and Kidney Institute, Cleveland, Ohio
  - Basel Hassoun, Oklahoma City, Oklahoma
  - Michael England, MD, Texas Health Care, Fort Worth, Texas
  - Michael DeBakey VA Med Ctr, Houston, Texas
- Canada (4):
  - Northern Alberta Urology Center, Edmonton, Alberta
  - Silverado Research, Inc, Victoria, British Columbia
  - Toronto Western Hospital, Toronto, Ontario
  - University of Sherbrooke, Sherbrooke, Quebec

IPD SHARING:
Plan to Share IPD: No